CLINICAL TRIAL: NCT06373367
Title: Preeclampsia Educational Program Study
Brief Title: Preeclampsia Educational Program Study (PrEPS)
Acronym: PrEPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Principal Investigator, Megan Oakes, MD MCSI, MemorialCare Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 461-24
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Preeclampsia; Preeclampsia Severe; Preeclampsia Mild; Preeclampsia Postpartum
Keywords: preeclampsia; education
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Illustration (Experimental): This study arm will receive education via an illustration based application
  Interventions: Other: Illustration based application
- Text (Active Comparator): This study arm will receive education via text based application
  Interventions: Other: Text based application

INTERVENTIONS:
Other: Illustration based application — Illustrations regarding the cause, risks, and warning signs of preeclampsia
  Arms: Illustration
Other: Text based application — Standard preeclampsia discharge instructions
  Arms: Text

SUMMARY:
Preeclampsia complicates approximately 8% of all pregnancies. A critical factor of outpatient monitoring is patient education; specifically, education regarding nature of the disease, ongoing short- and long-term risks, and warning signs and symptoms for worsening of disease. This study aims to compare patient knowledge using a novel illustration based app compared to standard discharge instructions.

DETAILED DESCRIPTION:
Preeclampsia complicates approximately 8% of all pregnancies. While many patients improve following delivery, the disease process remains a leading cause for postpartum morbidity and mortality. A critical factor of outpatient monitoring is patient education; specifically, education regarding nature of the disease, ongoing short- and long-term risks, and warning signs and symptoms for worsening of disease. There is a gap in the literature regarding effective, patient-centered educational tools specifically addressing these elements, especially in the postpartum period.

The investigators propose a pilot, randomized controlled trial of postpartum patients with preeclampsia. The intervention of interest is an illustration-based, educational mobile device application (app) focused on the short- and long-term risks associated with preeclampsia and warning signs and symptoms of worsening disease postpartum. The control for this study will be the same information in a text-only format, also accessed through a mobile device app.

The investigators central hypothesis is that an illustration-based app will improve knowledge of preeclampsia among postpartum patients compared to text-only educational material.

Specific Aim 1: Compare the difference in preeclampsia knowledge score from text-only versus illustration-based education 24 hours post intervention (short-term). The investigators hypothesize that patients who receive illustration-based education will have a) higher preeclampsia knowledge scores at 24 hours post-intervention compared to text-only educational materials and b) a greater increase in preeclampsia knowledge score from baseline (pre-test) compared to text-only education.

Specific Aim 2: Compare the difference in preeclampsia knowledge score from text-only versus illustration-based education >4 weeks post intervention (long-term). The investigators hypothesize that patients who receive illustration-based education will have a) higher preeclampsia knowledge scores at > 4 weeks post-intervention compared to text-only educational materials and b) a greater increase in preeclampsia knowledge score from baseline (pre-test) compared to text-only education.

ELIGIBILITY:
Inclusion Criteria:

* Preeclampsia with or without severe features
* Able to read and speak English
* Consistent access to mobile device with QR-reading capability and ability to access mobile-device application.
* Pre-and postnatal care provided by OB Clinic (resident clinic) or Magella (maternal-fetal medicine)

Exclusion Criteria:

* Patient age < 18 years old
* Non-English speaking
* Current enrollment in another trial targeting postpartum preeclampsia parameters
* Arm width >40cm (XL Cuff)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia knowledge score - short | Measured at 24 hours postpartum
  Short term preeclampsia knowledge score. Scored from 0-24, with 24 demonstrating the most correct answers to the assessment

SECONDARY OUTCOMES:
Preeclampsia knowledge score - long | Measured between 4 - 6 weeks postpartum
  Long term preeclampsia knowledge score. Scored from 0-24, with 24 demonstrating the most correct answers to the assessment
GAD-7 score | Measured between 4-6 weeks postpartum
  Generalized anxiety score. A score of 0-4 demonstrating none or minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, 15-21 severe anxiety
72 hour BP check | Measured 72 hours after hospital discharge
  Adherence to a blood pressure check
Number of participants who attend a postpartum visit | Measured within 6 weeks postpartum
  Adherence to one postpartum visit
Daily BP recordings | Measured within 6 weeks postpartum
  Percent of daily blood pressure recordings at home
Accessed material | Measured at 6 weeks postpartum
  Number of times information accessed postpartum
Unplanned readmission | Measured at 6 weeks postpartum
  Number of unplanned readmissions related to preeclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Megan Oakes, MD MSCI, Principal Investigator — Magella Medical Group, MemorialCare
Locations (1):
- MemorialCare Long Beach Medical Center, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Igdoura SA, Herscovics A, Lal A, Moremen KW, Morales CR, Hermo L. Alpha-mannosidases involved in N-glycan processing show cell specificity and distinct subcompartmentalization within the Golgi apparatus of cells in the testis and epididymis. Eur J Cell Biol. 1999 Jul;78(7):441-52. doi: 10.1016/s0171-9335(99)80071-5. PMID 10472797
- [Background] Dol J, Hughes B, Bonet M, Dorey R, Dorling J, Grant A, Langlois EV, Monaghan J, Ollivier R, Parker R, Roos N, Scott H, Shin HD, Curran J. Timing of maternal mortality and severe morbidity during the postpartum period: a systematic review. JBI Evid Synth. 2022 Sep 1;20(9):2119-2194. doi: 10.11124/JBIES-20-00578. PMID 35916004
- [Background] Shree R, Hatfield-Timajchy K, Brewer A, Tsigas E, Vidler M. Information needs and experiences from pregnancies complicated by hypertensive disorders: a qualitative analysis of narrative responses. BMC Pregnancy Childbirth. 2021 Nov 2;21(1):743. doi: 10.1186/s12884-021-04219-0. PMID 34724906
- [Background] You WB, Wolf MS, Bailey SC, Grobman WA. Improving patient understanding of preeclampsia: a randomized controlled trial. Am J Obstet Gynecol. 2012 May;206(5):431.e1-5. doi: 10.1016/j.ajog.2012.03.006. Epub 2012 Mar 13. PMID 22542120
- [Background] You WB, Wolf M, Bailey SC, Pandit AU, Waite KR, Sobel RM, Grobman W. Factors associated with patient understanding of preeclampsia. Hypertens Pregnancy. 2012;31(3):341-9. doi: 10.3109/10641955.2010.507851. Epub 2010 Sep 22. PMID 20860492
- [Background] Chames MC, Livingston JC, Ivester TS, Barton JR, Sibai BM. Late postpartum eclampsia: a preventable disease? Am J Obstet Gynecol. 2002 Jun;186(6):1174-7. doi: 10.1067/mob.2002.123824. PMID 12066093
- [Background] Collier AY, Molina RL. Maternal Mortality in the United States: Updates on Trends, Causes, and Solutions. Neoreviews. 2019 Oct;20(10):e561-e574. doi: 10.1542/neo.20-10-e561. PMID 31575778
- [Background] Ditisheim A, Wuerzner G, Ponte B, Vial Y, Irion O, Burnier M, Boulvain M, Pechere-Bertschi A. Prevalence of Hypertensive Phenotypes After Preeclampsia: A Prospective Cohort Study. Hypertension. 2018 Jan;71(1):103-109. doi: 10.1161/HYPERTENSIONAHA.117.09799. Epub 2017 Nov 13. PMID 29133363
- [Background] Gestational Hypertension and Preeclampsia: ACOG Practice Bulletin, Number 222. Obstet Gynecol. 2020 Jun;135(6):e237-e260. doi: 10.1097/AOG.0000000000003891. PMID 32443079